CLINICAL TRIAL: NCT02840032
Title: Role of Ultrasonography in the Diagnosis of Pneumothorax Following Transbronchial Biopsy in LungTransplant Patients.
Brief Title: Determination of Pneumothorax Post Lung Biopsy
Status: Withdrawn | Type: Observational
Why Stopped: No subjects enrolled
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: 1606M88672
Record Dates: First submitted 2016-07-18; First posted 2016-07-21 (Estimated); Last update posted 2018-05-03 (Actual); Status verified 2018-04

CONDITIONS: Pneumothorax
MeSH Terms: conditions — Pneumothorax

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Bedside ultrasonography for detection of pneumothorax after transbronchial lung biopsies in lung transplant patients

DETAILED DESCRIPTION:
The patients who undergo transbronchial forceps lung biopsies get a routine CXR after the biopsies are performed. The reason for CXR is to find out if pneumothorax occurred or not. CXR is required patient transportation and interpretation by the radiologist as well as time consuming. Instead, we are planning to perform bedside ultrasound to determine if pneumothorax occurred or not

ELIGIBILITY:
Inclusion Criteria:

* Any lung transplant patient who undergoes to bronchoscopic lung biopsy

Exclusion Criteria:

* Patients develop respiratory failure during the procedure

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Lung transplant patients who undergo routine bronchoscopic biopsy procedure for rejection determination
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2016-07; Primary Completion 2017-08 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
Determination of pneumothorax after transbronchial lung biopsy | 2 hours

CONTACTS AND LOCATIONS:
Overall Officials: Erhan Dincer, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Undecided